CLINICAL TRIAL: NCT05245331
Title: High-volume and Low-volume Water Transanal Irrigation for the Management of Low Anterior Resection Syndrome. A Crossover Randomized Controlled Clinical Trial.
Brief Title: Transanal Irrigation for Low Anterior Resection Syndrome.
Acronym: HiLoV_TAI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Asociacion Española de Coloproctologia (Other); Asociación Española de Cirugía (Unknown)
Responsible Party: Principal Investigator, Loris Trenti, Principal Investigator, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PR297/21
Record Dates: First submitted 2022-01-07; First posted 2022-02-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Low Anterior Resection Syndrome
Keywords: Rectal Cancer; LARS; Low Anterior Resection Syndrome; Transanal Irrigation
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-volume TAI (Active Comparator): This group will be instructed on High-volume TAI to be perform daily or every 2 days for 2 months. After 15 days of wash-out they will switch to Low-TAI treatment for 2 months.
  Interventions: Device: Peristeen® Transanal irrigation system with the conic catheter; Device: Standard reusable enema
- Low volume - TAI (Active Comparator): This group will be instructed on Low-volume TAI to be perform daily or every 2 days for 2 months. After 15 days of wash-out they will switch to the Low-TAI treatment for 2 months.
  Interventions: Device: Peristeen® Transanal irrigation system with the conic catheter; Device: Standard reusable enema

INTERVENTIONS:
Device: Peristeen® Transanal irrigation system with the conic catheter — The High-TAI (400-1000ml) will be self-performed using the Peristeen® Transanal irrigation system with the conic catheter every 48 hours during the first two week of treatment. Then patients could change frequency and volume of TAI depending on their needs and/or preference.
  The Low-TAI will be self-performed using a standard 250ml water enema every 48 hours during the first two week of treatment. Then patients could change frequency of TAI depending on their needs and/or preference.
Device: Standard reusable enema — The High-TAI (400-1000ml) will be self-performed using the Peristeen® Transanal irrigation system with the conic catheter every 48 hours during the first two week of treatment. Then patients could change frequency and volume of TAI depending on their needs and/or preference.
  The Low-TAI will be self-performed using a standard 250ml water enema every 48 hours during the first two week of treatment. Then patients could change frequency of TAI depending on their needs and/or preference.

SUMMARY:
The aim of this study is to investigate whether the high-volume transanal irrigation (TAI) performed by the Peristeen Plus® system is superior to the low-volume TAI performed by standard 250ml water enema for the treatment of Low Anterior Resection Syndrome (LARS).

DETAILED DESCRIPTION:
Most of the patients operated on for rectal cancer present defecatory disfunction symptoms known as Low Anterior Resection Syndrome (LARS) of different degree and severity. Although, transanal irrigation (TAI) has been shown to be useful in improve LARS and quality of life of these patients no evidence exists about the best way to realize TAI in terms of irrigation volume and systems and frequency of irrigation. This crossover randomized controlled trial aims to evaluate the impact of two different type of TAI (high-volume by Peristeen Plus® and low-volume performed by 250ml water enema) on LARS and quality of life in patients with major LARS secondary to low anterior rectal resection (LAR) for primary rectal cancer. The primary outcome is the reduction of LARS score after two months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Personal history of LAR or ultra-LAR with total mesorectal excision (TME) and sphincter preservation with stapled or manual end to end anastomosis for primary rectal cancer.
* Major LARS (score 30-42).
* At least 1 year follow-up after LAR or ultra-LAR or temporary stoma closure.
* Anastomotic integrity demonstrated by endoscopic, radiologic or clinical examination.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) between 0-2.
* Age≥ 18 years

Exclusion Criteria:

* Side to end mechanical anastomosis or J-pouch colorectal anastomosis
* Partial or total intersphincteric resection.
* Personal history of anastomotic dehiscence, chronic pelvic sepsis, anastomotic sinus, anastomotic stricture or other any other anastomotic complications.
* Persona history of other colorectal, proctologic or pelvis surgery or disease.
* Personal history of bariatric surgery.
* Functioning sacral neurostimulator carriers.
* Previous use of transanal irrigation systems for LARS treatment
* Presence of an ostomy.
* Local or distant rectal cancer recurrence and/or any other active neoplastic disease.
* Altered cognitive status.
* Pregnancy and age < 18 years
* Any other diseases that may alter results of the study.
* Refusal to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
LARS score | day 1st, 30th, 60th, 75th, 105th, and 135th.
  LARS score changes with treatments.
  No LARS: 0-20; Minor LARS 21-29; Major LARS 30-42.

SECONDARY OUTCOMES:
Daily bowel movements number (total, day, and night) | recorded daylily during the last 15 days at basal time and at day 60th, 75th, and 135th)
  Defecation habits change with treatments
Short Form 36 quality of live questionnaire (SF-36) | day 1st, 30th, 60th, 75th, 105th, and 135th.
  Quality of life changes with treatments.
  Values between 0-100 (higher score means better outcome).
Vaizey score | day 1st, 30th, 60th, 75th, 105th, and 135th.
  Fecal incontinence symptoms change with treatments.
  Values between 0-24 (higher score means worse outcome).
Satisfaction grade (VAS: 0-10). | day 1st, 30th, 60th, 75th, 105th, and 135th.
  Patients' satisfaction grade related with treatments
Preferred treatments | day 135
  What treatment is preferred by the patients after having tried both
Adverse effects related to both treatments. | day 1 to 135.
  Adverse effects and complication directly related with one of the two treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Loris Trenti, PhD, Principal Investigator
Locations (2):
- Spain (2):
  - Bellvitge University Hospital, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona

IPD SHARING:
Plan to Share IPD: No